CLINICAL TRIAL: NCT06955260
Title: A Randomized Trial of SGLT2 Inhibition With Empagliflozin in Adults With Fontan Circulatory Failure (EMPA-HEART 3 CardioLink-12)
Brief Title: SGLT2 Inhibition With Empagliflozin in Fontan Circulatory Failure
Acronym: EMPA-HEART-3
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Subodh Verma (Other)
Collaborators: Boehringer Ingelheim (Industry); Applied Health Research Centre (Other)
Responsible Party: Sponsor-Investigator, Subodh Verma, Professor of Surgery and Pharmacology & Toxicology, Canadian Medical and Surgical Knowledge Translation Research Group
Organization: Canadian Medical and Surgical Knowledge Translation Research Group (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1245-0331
Record Dates: First submitted 2025-03-15; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Congenital Heart Disease
Keywords: Fontan Circulatory Failure; Empagliflozin; Double-blind; randomized
MeSH Terms: conditions — Heart Defects, Congenital | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized (1:1), placebo-controlled, parallel group trial of empagliflozin vs. placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin (Active Comparator)
  Interventions: Drug: Empagliflozin 10 mg
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Empagliflozin 10 mg — Participants will take 10 mg of empagliflozin once daily
  Arms: Empagliflozin
Other: Placebo — Participants will take 10 mg of placebo once daily
  Arms: Placebo

SUMMARY:
Some people are born with a birth defect where they only have one functioning ventricle (lower chamber) in their heart. This condition can be initially managed with a Fontan operation, but there is a risk of developing Fontan Circulatory Failure (FCF) later in life. FCF occurs when the single working heart ventricle is no longer strong enough to pump blood throughout the body. This also means the heart has difficulty supplying oxygen to keep up with the needs of the body. As a result, individuals living with FCF may have some challenges carrying out day to day activities. A heart transplant is currently the only therapeutic option for individuals living with FCF. The investigators are conducting this trial to determine whether a medication called empagliflozin can help these people have a better quality of life.

DETAILED DESCRIPTION:
EMPA-HEART 3 CardioLink-12 is a global, multicentre, randomized, double-blinded, placebo-controlled, parallel group trial of empagliflozin vs. placebo in addition to standard of care therapy in adults with Fontan Circulatory Failure (FCF). A total of 410 individuals who provide written informed consent and meet the inclusion criteria following screening will be randomized (1:1) to receive either empagliflozin 10 mg once daily or matching placebo. During the 12-week follow-up, there will be four in-person and three telephone/virtual assessment visits.

The primary goal of this investigation is to determine whether 12 weeks of therapy with the sodium-glucose cotransporter 2 (SGLT2) inhibitor, empagliflozin, will improve clinical and participant-reported outcome measures in adults with FCF.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years of age) with FCF, defined by dysfunction of the Fontan physiology that causes limitation to the individual's ability to carry out daily life activities, on standard of care therapy

Exclusion Criteria:

* Diuretic initiation or dose change ≤2 weeks prior to enrollment On a SGLT2 inhibitor currently or within 12-weeks prior to enrollment in the trial
* Allergic to or has a known intolerance to any of the ingredients in empagliflozin or other SGLT2 inhibitors
* Pregnant or planning a pregnancy during the duration of the trial or breast feeding
* Living with type 1 diabetes mellitus
* Has an unresolved acute illness (e.g., acute appendicitis, COVID-19, gastroenteritis)
* History of ketoacidosis
* Has an estimated glomerular filtration rate (eGFR) that is <30 mL/min/1.73 m2 Total bilirubin, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥2-fold upper limit of normal (ULN) at screening
* Has a baseline systolic BP that is <80 mmHg or ≥200 mmHg
* Planned hospital intervention during trial period for management of FCF defined as one of the following:
* Admission for intravenous diuretics
* Admission for intravenous inotropes
* Admission for ascites drainage
* Admission for new or worsening ascites of clinical significance
* Admission for management of arrhythmia
* Admission for management of lymphatic dysfunction
* Admission for interventional cardiological or cardiac surgical procedure within 30-days prior to screening, or consideration for any cardiac surgical or interventional cardiological procedure during trial participation
* Admission for cardiac resynchronization therapy within 90-days prior to screening, or consideration of cardiac resynchronization therapy during trial participation
* Is unable to provide written informed consent, complete the trial or comply with the requirements of the trial protocol
* Participation in other interventional studies within 30-days of the screening visit that could influence any of the trial outcomes (exclusive of observational registries)
* Received intravenous diuretic within the previous 14-days
* On a heart transplant waiting list
* Current or imminent hospitalization for management of FCF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Hierarchical endpoint | Week 12
  Primary hierarchical composite outcome will be analyzed using a win ratio based on the Finkelstein-Schoenfeld test.
  * All cause death (no. of participants)
  * Listing for heart transplantation or initiation of mechanical circulatory support (no. of participants)
  * Sustained ventricular tachycardia or aborted sudden cardiac death (no. of participants)
  * Hospital admission for management of FCF defined by any of the following:
    * Admission for intravenous diuretics (no. of participants)
    * Admission for intravenous inotropes (no. of participants)
    * Admission for ascites drainage (no. of participants)
    * Admission for management of new or worsening ascites of clinical significance (no. of participants)
    * Admission for management of arrhythmia (no. of participants)
    * Admission for management of lymphatic dysfunction (no. of participants)
  * ≥5 points change in the KCCQ-Clinical Summary Score (KCCQ-CSS) from baseline to Week 12
  * Change in 6-minute walk distance f

SECONDARY OUTCOMES:
All cause death | Week 12
  All cause death (no. of participants)
Listing for heart transplantation or initiation of mechanical circulatory support | Week 12
  Listing for heart transplantation or initiation of mechanical circulatory support (no. of participants)
Sustained ventricular tachycardia or aborted sudden cardiac death | Week 12
  Sustained ventricular tachycardia or aborted sudden cardiac death (no. of participants)
Hospital admission for management of FCF | Week 12
  Hospital admission for management of FCF (in number of participants) as defined by any of the following:
  * Admission for intravenous diuretics (no. of participants)
  * Admission for intravenous inotropes (no. of participants)
  * Admission for ascites drainage (no. of participants)
  * Admission for management of new or worsening ascites of clinical significance (no. of participants)
  * Admission for management of arrhythmia (no. of participants)
  * Admission for management of lymphatic dysfunction (no. of participants)
Change in KCCQ-Clinical Summary Score | Week 12
  ≥5 points change in the KCCQ-Clinical Summary Score (KCCQ-CSS) from baseline (no. of participants)
Change in 6-minute walk test | Week 12
  Change in 6-minute walk distance (in meters)
Time to severe FCF | Week 12
  Time to severe FCF, defined as the first occurrence of any of the following:
  * Death (days)
  * Placement on heart or combined heart and liver transplantation list (days)
  * Initiation of palliative care because the individual is not a heart transplant candidate (days)
  * Fontan take down surgery (days)
Change in FCF status | Week 12
  Investigator-reported global change in FCF status (days)

OTHER OUTCOMES:
Fontan revision surgery | Week 12
  Time to Fontan revision surgery: atrioventricular valve replacement or repair, aortic valve replacement, Fontan conduit replacement (days)
Fontan conversion surgery | Week 12
  Time to Fontan conversion surgery from right atrial-pulmonary artery to lateral tunnel or extracardiac (days)
Change in cardiopulmonary exercise testing (CPET) variables if collected for clinical reasons | Week 12
  Blood pressure (BP) at baseline and peak exercise (mmHg)
Change in cardiopulmonary exercise testing (CPET) variables if collected for clinical reasons | Week 12
  Heart rate at baseline and peak exercise (BPM)
Change in cardiopulmonary exercise testing (CPET) variables if collected for clinical reasons | Week 12
  Peak oxygen consumption (VO2) in mL/kg/min
Change in cardiopulmonary exercise testing (CPET) variables if collected for clinical reasons | Week 12
  Peak oxygen consumption (VO2) as % of predicted
Change in cardiopulmonary exercise testing (CPET) variables if collected for clinical reasons | Week 12
  VO2 at anaerobic threshold in mL/kg/min
Change in cardiopulmonary exercise testing (CPET) variables if collected for clinical reasons | Week 12
  VO2 at anaerobic threshold as % of predicted
Change in cardiopulmonary exercise testing (CPET) variables if collected for clinical reasons | Week 12
  Ventilatory efficiency (VE)/volume of carbon dioxide produced (VCO2) ratio at anaerobic threshold and at peak exercise
Change in cardiopulmonary exercise testing (CPET) variables if collected for clinical reasons | Week 12
  O2 pulse at peak exercise (% predicted)
Change in cardiopulmonary exercise testing (CPET) variables if collected for clinical reasons | Week 12
  Time of exercise (min)
Change in cardiopulmonary exercise testing (CPET) variables if collected for clinical reasons | Week 12
  Load of exercise (in Watts if measured on bike, or in metabolic equivalents [METs] if measured on treadmill)
Change in cardiopulmonary exercise testing (CPET) variables if collected for clinical reasons | Week 12
  Ventilation (VE) at peak exercise in L/min
Change in cardiopulmonary exercise testing (CPET) variables if collected for clinical reasons | Week 12
  Forced expiratory volume in 1 second (FEV1) in L
Change in cardiopulmonary exercise testing (CPET) variables if collected for clinical reasons | Week 12
  Forced vital capacity (FVC) in L
NT-proBNP | Week 12
  Change in N-terminal pro-B-type natriuretic peptide (pg/mL)
Hemoglobin | Week 12
  Change in hemoglobin (g/L)
Change in KCCQ score | Week 12
  Change in Kansas City Cardiomyopathy Questionnaire (KCCQ)-Overall Summary Score (KCCQ-OSS) and KCCQ-Total Summary Score (KCCQ-TSS) of ≥5 points. The KCCQ is scored on a scale from 0-100, with higher scores indicative of better health status.
Absolute change in KCCQ score | Week 12
  Absolute change in Kansas City Cardiomyopathy Questionnaire (KCCQ)-Clinical Score Summary (KCCQ-CSS), KCCQ-Overall Summary Score (KCCQ-OSS) and KCCQ-Total Summary Score (KCCQ-TSS). The KCCQ is scored on a scale from 0-100, with higher scores indicative of better health status.

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No